CLINICAL TRIAL: NCT03269448
Title: Correlation Between Peripheral and Central Venous Blood Partial Pressure of Carbon Dioxide in Critical Ill Patients
Status: Completed | Type: Observational
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Thanist Pravitharangul, MD, Ramathibodi Hospital
Other Study IDs: 011674
Record Dates: First submitted 2017-08-28; First posted 2017-08-31 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Partial Pressure of Carbon Dioxide
Keywords: partial pressure of carbon dioxide; carbon dioxide; peripheral venous blood; central venous blood; venous blood gas; blood gas analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Peripheral venous blood sampling — Blood collected from peripheral venous (extremities) and central venous (central catheter) for blood gas analyses
  Other Names: Central venous blood sampling

SUMMARY:
Observational study to analyze correlation between partial pressure of carbon dioxide from blood obtained from peripheral and central veins

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to institutional ICU with central venous catheter in place
* Venous blood gas analysis ordered

Exclusion Criteria:

* Central venous catheter malposition
* Difficult peripheral venous access

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admiited to institutional ICU with central venous catheter in place
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-03-10 (Actual); Study Completion 2018-03-10 (Actual)

PRIMARY OUTCOMES:
Difference between partial pressure of carbon dioxide | 30 minutes
  Difference between partial pressure of carbon dioxide taken from peripheral and central veins

CONTACTS AND LOCATIONS:
Overall Officials: Thanist Pravitharangul, MD, Study Chair — Ramathibodi Hospital
Locations (1):
- Department of Anesthesiology, Ramathibodi Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No